CLINICAL TRIAL: NCT01045070
Title: Periodontitis and Its Microbiological Agents as Prognostic Factors in Patients With Coronary Heart Disease
Brief Title: Periodontitis and Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: The German Heart Foundation (Other)
Responsible Party: Principal Investigator, Axel Schlitt, PD Dr. med. habil., Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: F/34/08
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Periodontitis; Coronary Heart Disease
Keywords: periodontitis and coronary heart disease
MeSH Terms: conditions — Periodontitis; Coronary Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood-samples and samples from gingival pockets
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- coronary heart disease

SUMMARY:
"Atherosclerosis is an inflammatory disease". The hypothesis of an infectious burden as trigger or initiator of the inflammatory process in atherosclerosis has been extensively discussed in the past years. One part of this discussion is focused on the infectious agents responsible for periodontitis. Several studies have found an association of periodontitis and/or bacteria related to this disease and atherosclerosis. However, a study focussing on the prognostic relevance of these factors is missing.

The hypothesis of this study is that periodontitis is a prognostic relevant risk factor for patients with angiographically proven coronary heart disease. Furthermore, the infectious pathogen burden by PCR-detection of periodontal pathogens will be evaluated as a prognostic factor.

960 consecutive patients with angiographically proven coronary heart disease will be included in this study. After inclusion of patients an extensive periodontal examination including PCR-sampling for 11 bacteria (Porphyromonas gingivitis, Actinobacillus actinomycetemcomitans, and others) will be performed. After 12 months patient will be follow up for any major adverse events (cardiovascular death, myocardial infarction, stroke).

If this study will find a relation of periodontitis or its microbiological agents to cardiovascular outcome of patients with coronary heart disease, further studies are necessary to investigate potential therapeutic consequences for patients with CHD and periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Coronary heart disease as defined by previous or current detection of 50% stenosis of a main coronary artery by coronary angiography or previous or current percutaneous coronary intervention (PCI) or previous or current coronary artery bypass surgery (CABG)

Exclusion Criteria:

* Inability to give written informed consent
* Periodontal treatment and/or antibiotic therapy during the last 6 months
* Pregnancy
* Current alcohol or drug abuse, or psychological reasons that make study participation impractical
* Drugs which are potential causal for gingival hyperplasia (Hydantoin, Nifedipine, Cyclosporin A, and other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary heart disease, admitted to the Martin Luther-University Halle-Wittenberg
Sampling Method: Probability Sample
Enrollment: 960 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Combined endpoint: myocardial infarction, cardiovascular death, stroke | 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Axel Schlitt, MD, Principal Investigator — Department of Medicine III, Martin Luther-University Halle-Wittenberg
Locations (1):
- Martin Luther-University Halle-Wittenberg, Halle, Germany

REFERENCES:
- [Derived] Reichert S, Rehm S, Schlitt A, Schulz S. Severe Periodontitis is Associated With Recurrent Cardiovascular Events-A 10-Year Longitudinal Cohort Study. J Periodontal Res. 2025 Dec;60(12):1201-1211. doi: 10.1111/jre.13365. Epub 2024 Nov 22. PMID 39578376
- [Derived] Schulz S, Rehm S, Schlitt A, Bitter K, Reichert S. The Interleukin 6 Protein Level as well as a Genetic Variants, (rs1800795, rs1800797) Are Associated with Adverse Cardiovascular Outcomes within 10-Years Follow-Up. Cells. 2023 Nov 28;12(23):2722. doi: 10.3390/cells12232722. PMID 38067150
- [Derived] Schulz S, Rehm S, Schlitt A, Lierath M, Ludike H, Hofmann B, Bitter K, Reichert S. C-Reactive Protein Level and the Genetic Variant rs1130864 in the CRP Gene as Prognostic Factors for 10-Year Cardiovascular Outcome. Cells. 2023 Jul 4;12(13):1775. doi: 10.3390/cells12131775. PMID 37443809
- [Derived] Schulz S, Zielske M, Schneider S, Hofmann B, Schaller HG, Schlitt A, Reichert S. Polymorphism of CD14 Gene Is Associated with Adverse Outcome among Patients Suffering from Cardiovascular Disease. Mediators Inflamm. 2021 Jul 8;2021:3002439. doi: 10.1155/2021/3002439. eCollection 2021. PMID 34305452
- [Derived] Reichert S, Seitter L, Schaller HG, Schlitt A, Schulz S. ANRIL polymorphisms (rs1333049 and rs3217992) in relation to plasma CRP levels among in-patients with CHD. Cytokine. 2020 Mar;127:154932. doi: 10.1016/j.cyto.2019.154932. Epub 2019 Nov 27. PMID 31770616
- [Derived] Schulz S, Schlitt A, Hofmann B, Schaller HG, Reichert S. Periodontal pathogens and their role in cardiovascular outcome. J Clin Periodontol. 2020 Feb;47(2):173-181. doi: 10.1111/jcpe.13224. Epub 2019 Dec 16. PMID 31765020
- [Derived] Reichert S, Schlitt A, Benten AC, Hofmann B, Schaller HG, Schulz S. Data on IL-6 c.-174 G>C genotype and allele frequencies in patients with coronary heart disease in dependence of cardiovascular outcome. Data Brief. 2016 Jul 16;8:1295-9. doi: 10.1016/j.dib.2016.07.020. eCollection 2016 Sep. PMID 27570807
- [Derived] Schulz S, Schlitt A, Lutze A, Lischewski S, Seifert T, Dudakliewa T, Gawe R, Werdan K, Hofmann B, Glaser C, Schaller HG, Reichert S. The importance of genetic variants in TNFalpha for periodontal disease in a cohort of coronary patients. J Clin Periodontol. 2012 Aug;39(8):699-706. doi: 10.1111/j.1600-051X.2012.01909.x. Epub 2012 Jun 12. PMID 22691114